CLINICAL TRIAL: NCT07234994
Title: Effect of Ozonized Gel Compared to Photobiomodulation Therapy on Wound Healing Following Surgical Gingivectomy : A Randomized Controlled Clinical Trial
Brief Title: Comparison of the Effect of Ozonized Gel to That of Photobiomodulation Therapy on Wound Healing Following Surgical Gingivectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mennatullah osama ahmed zaki wahba (Other)
Responsible Party: Sponsor-Investigator, Mennatullah osama ahmed zaki wahba, Dentist, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9245845
Record Dates: First submitted 2025-11-16; First posted 2025-11-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Gingival Enlargement
Keywords: Ozonized gel; Photobiomodulation Therapy; Surgical gingivectomy; Wound healing
MeSH Terms: conditions — Gingival Hyperplasia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ozonized gel group (Active Comparator): Application of ozonized gel to raw wound area following surgical gingivectomy.
  Interventions: Drug: ozonized gel application
- Photobiomodulation therapy group (Active Comparator): Application of diode laser 635nm to wound area following surgical gingivectomy
  Interventions: Device: photobiomodulation therapy using diode laser
- Control group (No Intervention): Spontaneous healing of wound area following surgical gingivectomy

INTERVENTIONS:
Drug: ozonized gel application — Application of ozonized gel to raw wound area following surgical gingivectomy.
  Arms: Ozonized gel group
Device: photobiomodulation therapy using diode laser — Application of diode laser 635nm to wound area following surgical gingivectomy
  Arms: Photobiomodulation therapy group

SUMMARY:
The goal of this clinical trial is to compare the effect of photobiomodulation to ozonized gel on wound healing following gingivectomy procedure on adults. The main questions it aims to answer are:

Which treatment modality provides less painful and more efficient wound healing ? What are the patient's feedback on different treatment modalities ? Researchers will compare ozonized gel to photobiomodulation to normal gingivectomy procedure with no interference.

Participants will:

Receive either ozonized gel or photobiomodualtion treatment following surgical gingivectomy Visit the clinic every 3,7,14 and 28 days for checkups and investigations

DETAILED DESCRIPTION:
Surgical gingivectomy is performed for elimination of supra bony pockets and gingival enlargements and it can be considered the gold standard treatment for such cases. The healing of wound site after gingivectomy occurs slowly by secondary intention; therefore, several studies have been conducted evaluating the effect of various treatment modalities to accelerate the process of wound healing such as use of ozonized gel and photobiomodulation. Ozone, owing to its biocompatibility, healing, and antimicrobial properties, is used for wound healing and tissue repair. Photobiomodulation Therapy (PBMT) using diode laser is another treatment modality regarded as an effective modality for the repair of tissues, control of pain and wound healing. This study will be carried out to clinically compare and evaluate the healing of surgical gingivectomy wounds using ozonized gel and PBMT.

Aim: Compare the efficacy of the ozonized gel to photobiomodulation therapy in wound healing following surgical gingivectomy Materials and Methods: This randomized controlled clinical trial will involve 48 surgical gingivectomy wound sites, equally divided into three groups, Group-I (test group1): ozonized hydrogel will be applied to raw wound area following surgical gingivectomy and at days 3,7,14 post surgery. Group II (test group 2): the surgical site will be irradiated with a diode laser (635 nm,50mW) directly following surgery and at days 3,7,14 postoperative. Group III (control group) will include surgical gingivectomies that will be left to heal spontaneously. Wound healing will be assessed using Landry's Healing index and by measuring degree of epithelialization, and pain level will be assessed using a Visual analog scale on the 3rd, 7th, 14th, and 28th days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients indicated for surgical gingivectomy.
2. Adequate amount of keratinized tissue.
3. Average age between 18-40 years.
4. Well-educated patients as post-operative instructions need to be followed precisely.
5. Good oral hygiene with a full mouth O'Leary plaque index of less than or equal to 10% and a full mouth Gingival Index of zero

Exclusion Criteria:

1. History of smoking.
2. Patients who have any known systemic disease that interfere with performance of surgical gingivectomy or periodontal wound healing.
3. Patients who have any previous adverse reactions to the products (or similar products) used in this study.
4. Pregnant women.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-16 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Healing index (HI) using Landry index | day 3,7,14,28 post surgical gingivectomy
  The healing index (HI) scores will be assessed on the basis of redness, presence of granulation tissues, bleeding, suppuration, and epithelialization.
Evaluation of epithelialization of the wound area | days 0,3,7,14,28 post surgical gingivectomy
  A plaque disclosing agent is used to measure wound area epithelialization by dying the abraded and deepithelialized areas on the gingiva on postoperative days 3,7,14 and 28. By using this solution, assessment of degree of epithelialization and wound healing is made easier. Wound surface epithelialization in the obtaining photographs will be evaluated using an Image-analyzing software. To ensure standardization, all photographs will taken by the same person with the same camera at the same angle.
Postoperative pain using the VAS | day 3, day 7, and day 14 post surgery.
  Visual Analogue Scale (VAS) is a simple measurement tool that measures the intensity of pain as recorded by the patient. 10-point visual analog scale of pain rating, with 0 marked as "no pain" and 10 marked as "worst pain imaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt